CLINICAL TRIAL: NCT06974734
Title: AN OPEN-LABEL PHASE 1 STUDY TO EVALUATE PF-08046037 AS MONOTHERAPY AND PART OF COMBINATION THERAPY IN PARTICIPANTS WITH ADVANCED MALIGNANCIES
Brief Title: A Clinical Trial of PF-08046037 Alone or With Sasanlimab in Patients With Advanced or Metastatic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5941001; 2025-521499-69-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-22; First posted 2025-05-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non Small Cell Lung; Carcinoma, Pancreatic Ductal; Malignant Melanoma; Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Keywords: Advanced solid tumors; NSCLC; PDAC; HNSCC; ISAC; ADC; PD-L1 inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Pancreatic Ductal; Melanoma; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1a (Experimental): PF-08046037 monotherapy dose escalation
  Interventions: Drug: PF-08046037
- Part 2a (Experimental): PF-08046037 monotherapy dose optimization
  Interventions: Drug: PF-08046037
- Part 3a (Experimental): PF-08046037 monotherapy dose expansion
  Interventions: Drug: PF-08046037
- Part 1b (Experimental): PF-08046037 +sasanlimab dose escalation
  Interventions: Drug: PF-08046037; Drug: sasanlimab
- Part 2b (Experimental): PF-08046037 + sasanlimab dose optimization
  Interventions: Drug: PF-08046037; Drug: sasanlimab
- Part 3b (Experimental): PF-08046037 + sasanlimab dose expansion
  Interventions: Drug: PF-08046037; Drug: sasanlimab

INTERVENTIONS:
Drug: PF-08046037 — Given into the vein (IV; intravenous)
  Other Names: SGN-PDL1iT
Drug: sasanlimab — Given under the skin (SQ; subcutaneous)
  Other Names: PF-06801591
  Arms: Part 1b; Part 2b; Part 3b

SUMMARY:
The purpose of this study is to learn about the safety and the effects of PF-08046037 alone or with sasanlimab for the treatment of certain advanced or metastatic malignancies.

This study is seeking participants who:

* have advanced or metastatic non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), melanoma, or pancreatic ductal adenocarcinoma (PDAC);
* are able to provide tumor tissue samples;
* have measurable disease. All participants will receive while at the clinic PF-08046037 alone as an intravenous (IV) infusion (given directly into a vein) or with sasanlimab as a subcutaneous (SQ) injection (given under the skin) once every 3 weeks.

Participants will continue to take the study drug(s) until their cancer is no longer responding or if the patient cannot safely take them. The study team will monitor how each participant is doing with the study treatment during regular visits at the study clinic.

ELIGIBILITY:
This study is seeking participants who have the following tumor types and can provide tumor tissue samples as per below.

1. Tumor types

   * Monotherapy Dose Escalation (Part 1a) and Optimization (Part 2a) cohorts

     * Advanced or metastatic NSCLC, HNSCC, melanoma, or PDAC
     * Must have progressive disease following at least 1 prior approved systemic therapy
   * Monotherapy Dose Expansion (Part 3a)

     • Advanced or metastatic NSCLC or PDAC
   * Combination Safety Evaluation (Part 1b) and Dose Optimization (Part 2b)

     * Advanced or metastatic NSCLC or HNSCC
     * May be either a) not received prior immunotherapy for the tumor type OR b) relapse/ refractory after prior immunotherapy
   * Combination Dose Expansion (Part 3b)

     * Unresectable locally advanced or metastatic HNSCC or NSCLC
     * Must not have received prior systemic cytotoxic therapy in the locally advanced or metastatic setting (first-line setting)
     * Must be treatment naïve to any immunotherapy
     * NSCLC must have PD-L1 expression TPS >=50%
     * HNSCC must have PD-L1 expression CPS >=1
2. Tissue requirement

   * Part 1 at lower doses: sufficient archival tissue collected within 12 months of enrollment for submission to central laboratory
   * Part 1 at higher doses: de novo baseline tumor biopsy or archival tissue within 12 months of enrollment
   * Part 1 backfill: de novo baseline and on-treatment tumor biopsies are required
   * Part 2 and 3: de novo baseline or archival tissue within 6 months of enrollment
   * Part 2 and 3: mandatory on-treatment tumor biopsy, if required by sponsor
3. Measurable disease per RECIST v1.1

Participants who meet the following might not be able to participate.

1. History of Grade >=3 immune mediated AE related to prior immune modulatory therapy and required immunosuppressive therapy
2. Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent
3. History of uveitis within the preceding 6 months
4. Clinically significant Grade >=3 neurodegenerative disease
5. Grade 3 or higher pulmonary disease unrelated to underlying malignancy
6. Previous exposure to an investigational immunostimulatory antibody conjugate or systemic TLR agonist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days after the last study treatment, up to approximately 2 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of participants with laboratory abnormalities | Through 30-37 days after the last study treatment, up to approximately 2 years
Number of dose modifications due to AEs | Through end of treatment up to approximately 2 years
Number of participants with dose-limiting toxicities (DLTs) | Up to 21 days
Number of participants with DLTs by dose level | Up to 21 days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter - Area under the concentration-time curve (AUC) | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
PK parameter - Maximum concentration (Cmax) | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
PK parameter - Time to maximum concentration (Tmax) | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
PK parameter - t1/2 | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
PK parameter - Trough concentration (Ctrough) | Through 30-37 days after the last study treatment, up to approximately 2 years
  PK endpoint
Number of participants with antidrug antibodies (ADAs) | Through 30-37 days after the last study treatment, up to approximately 2 years
Objective response rate (ORR) | Through end of study and up to approximately 2 years
  The objective response rate (ORR) is defined as the percentage of participants with complete response (CR) or partial response (PR) which is subsequently confirmed as assessed according to Response Evaluation in Solid Tumors (RECIST) v1.1.
Best overall response | Through end of study and up to approximately 2 years
  The best overall response for a participant will be determined by the order of confirmed CR, confirmed PR, stable disease (SD), progressive disease (PD), not evaluable (NE) or not applicable (NA) per RECIST v1.1.
Duration of response (DOR) | Through end of study and up to approximately 2 years
  DOR is defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression per RECIST v1.1 or to death due to any cause
Progression-free survival (PFS) | Through end of study and up to approximately 2 years
  PFS is defined as the time from start of PF-08046037 to first documentation of disease progression (based on radiographic assessments per RECIST v1.1) or death due to any cause, whichever comes first
Overall survival (OS) | Through end of study and up to approximately 2 years
  OS is defined as the time from start of PF-08046037 to date of death due to any cause
Percent change of cells within tumors based on multiplex immunofluorescence | Through end of study and up to approximately 2 years
  This measure will assess the number of immune cells, PD-1, PD-L1, and TLR7 expression within the tumor microenvironment.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (17):
  - Presbyterian/ St. Lukes Medical Center, Denver, Colorado
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Smilow Cancer Hospital - Yale New Haven Health, New Haven, Connecticut
  - Yale - New Haven Hospital - Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - Smilow Cancer Hospital - Trumbull, Trumbull, Connecticut
  - Community Health Network, Inc, Indianapolis, Indiana
  - Community Health Network, Inc., Indianapolis, Indiana
  - START Midwest, Grand Rapids, Michigan
  - UPMC Vision Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Shadyside Hospital, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tristar Centennial Medical Center, Nashville, Tennessee
  - Methodist Hospital, San Antonio, Texas
  - START San Antonio, San Antonio, Texas
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5941001